CLINICAL TRIAL: NCT01933321
Title: Effect of Intrathecal Administration of Hematopoietic Stem Cells in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Chair of Hematology, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS and stem cell therapy
Record Dates: First submitted 2012-09-28; First posted 2013-09-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS, stem cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intrathecal autologous stem cells (Experimental): Intrathecal stem cells will be administered to patients that fulfill the inclusion criteria.
  Interventions: Biological: Intrathecal autologous stem cell

INTERVENTIONS:
Biological: Intrathecal autologous stem cell — Mobilization and collection of stem cells for intravenous and intrathecal administration

SUMMARY:
Autologous cell therapy in patients with ALS can stimulate neuroplasticity, modifying the neurodegenerative process and stops the clinical progression of disease.

DETAILED DESCRIPTION:
There is no more extensive information

ELIGIBILITY:
Inclusion Criteria:

* patients with a confirmed diagnosis of ALS according to El Escorial criteria. Diagnosis-time less than four years.
* Over 18 years old. Forced vital capacity ≥ 40%.
* One year of evolution.
* Adequate nutritional state

Exclusion Criteria:

* Severe bulbar ALS involucre.
* Inadequate nutritional status.
* Spondylotic myelopathy, or abnormalities in imaging study.
* Having concomitant neurological or psychiatric disease.
* Systemic disease with poor-control.
* History of treatment with steroids or immunoglobulins in the last year.
* Participate in the past three months in a Clinical Trial.
* History of malignancy or cancer today.
* Intracranial hypertension.
* Clinical suggestive data of infection in the site of lumbar puncture.
* Tracheostomy.
* Use of mechanical ventilation. Forced vital capacity less than 40%. HIV-seropositive or presence of antibodies against hepatitis B or C in the serological studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of autologous intrathecal administration of hematopoietic stem cells in patients with ALS. | up to 12 months

SECONDARY OUTCOMES:
To evaluate the safety of intrathecal administration of hematopoietic stem cells in patients with ALS. | During the procedure and at 1st, 2nd, 3rd, 6th and 12 th month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez-Almaguer, MD, Principal Investigator — Hospital Universitario "Dr. José Eleuterio González"; Jose C Jaime-Pérez, MD PhD, Study Director — Hospital Universitario "Dr. José Eleuterio González"; Héctor R Martínez-Rodríguez, MD PhD, Study Chair — Hospital Universitario "Dr. José Eleuterio González"
Locations (1):
- Servicio Hematología Hospital Universitario, Monterrey, Nuevo León, Mexico